CLINICAL TRIAL: NCT02255344
Title: Multicenter Study to Develop a Risk Model for Early Major Cardiovascular Events Based on the IMSS National Registry of Acute Coronary Syndromes (RENASCA IMSS). Stage 1
Brief Title: Multicenter Study to Develop a Risk Model for Early Major Cardiovascular Events
Acronym: RENASCA-IMSS
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Gabriela Borrayo Sanchez, Medical Programs Coordinator, Instituto Mexicano del Seguro Social
Other Study IDs: R-2014-785-051
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Risk Model; National Registry; Comprehensive Care Program; Major Cardiovascular Events
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ST-Elevation Myocardial Infarction: Consecutive patients of any gender between 18 and 90 years old, diagnosed with ST-Elevation Myocardial Infarction according to international diagnostic criteria - ACC / AHA / ESC, attended in representative hospitals of tertiary and secondary care in the IMSS will be studied
- Non ST Segment Elevation: Consecutive patients of any gender between 18 and 90 years old, diagnosed with Non ST Segment Elevation (NSTEMI/ Unstable angina) according to international diagnostic criteria - ACC / AHA / ESC, attended in representative hospitals of tertiary and secondary care in the IMSS will be studied

SUMMARY:
Through the National Registry of patients with ACS in the IMSS (RENASCA IMSS) the investigators will know the real world in terms of risk factors frequency, clinical presentation and its complications, and in the end they can build a risk model for early Major Cardiovascular Events (MACE).

DETAILED DESCRIPTION:
Introduction: Ischemic heart diseases as the leading cause of death in Mexico are mainly due to acute myocardial infarction. In this sense, reperfusion strategies are the cornerstone of treatment to reduce complications and costs; however, less than 50 percent of patients receive this treatment as a third of the world's population dies by this cause.

The World Health Organization (WHO) predicts for the next two decades about 23.5 million deaths worldwide by cardiovascular diseases. Particularly Acute Coronary Syndrome (ACS) caused in 2008 about seven million deaths worldwide. It is estimated that each year in Mexico around 300 thousand people suffer an ACS, at least 60 percent of these is caused by Myocardial Infarction (MI) but there are not real numbers for morbidity nor real clinical complications.

Efforts have been made in Mexican registries of ACS as shown in the first real world study done in the IMSS which serves the greater number of these cases (54.4 percent) called "National Registry of Acute Coronary Syndromes" (RENASCA IMSS). In this registry 10 tertiary care hospitals participated enrolling 2,398 patients with ACS diagnosis, most of them with ST-Elevation Myocardial Infarction (STEMI), representing 63 percent; the average age was 62 years. In 65 percent of cases stratified as high risk (GRACE> 150 points), only 42 percent were treated with fibrinolytic therapy, 8 percent with primary Percutaneous Coronary Intervention (PCI) and the remaining 50 percent did not receive any reperfusion therapy which is the cornerstone for the prognosis of these patients.

Currently Mexico is experiencing an increase in the elderly population and in the frequency of traditional risk factors for atherosclerosis associated with factors such as overweight and obesity which has become a high-risk population group for ischemic heart diseases and its complications. It represents a challenge to the health system from the point of view of prevention in the beginning but also in the diagnosis, prognosis, and treatment.

Treatment goals in traditional risk factors have not been accomplished yet. Patients are diagnosed late and there is not a risk model in our population since more than 50 percent of patients do not receive adequate treatment.

Therefore it is necessary to have a current outlook of what is happening in the mexican population through a National Registry of patients with ACS in the IMSS (RENASCA IMSS). This will allow to know the real world in terms of risk factors frequency, clinical presentation and its complications, and in the end a risk model can be built.

OBJECTIVE: To develop a risk model for early Major Cardiovascular Events (MACE) in patients with Acute Coronary Syndrome (ACS) based on the IMSS National Registry of Acute Coronary Syndromes (RENASCA IMSS.)

MATERIAL AND METHODS: Consecutive patients of any gender between 18 and 90 years old, diagnosed with Acute Coronary Syndrome (STEMI/ NSTEMI/ Unstable angina - according to international diagnostic criteria - American College of Cardiology (ACC) / American Heart Association (AHA) / European society of Cardiology (ESC), attended in representative hospitals of tertiary care in the IMSS will be studied.

The design is an analytical consecutive prospective multicenter study with an emerging cohort of patients with ACS through a National Registry in units of tertiary care in the IMSS (RENASCA IMSS). Follow-up will be done during hospitalization and 30 days, time of most Major Cardiovascular Events presentation (MACE) derived from the timing of initial treatment or lack of it.

MACE to evaluate during Follow-up will be: Reinfarction, myocardial ischemia, heart failure, electrocardiographic complications and / or death (mortality). 8 tertiary care hospitals or Medical Units of High Specialty (UMAES for its acronym in Spanish) will participated representing the country: an analysis of clinical and paraclinical variables contained in the record considered as relevant in predicting the inception cohort for MACE during hospitalization and 30 days will be done. The cohort of major cardiovascular events (as previously defined) will be compared with the cohort comprised by patients without such events.

Statistical analysis will be done with central tendency and dispersion measures according to the distribution of the variables. We will use the hypothesis testing according to the normality of data with T-test for independent groups or Mann-Whitney test for continuous variables, whereas for categorical variables X2 test or Fisher exact test when the observed frequency is <5 will be used. The free event will be analyzed with Kaplan Meier curves. To determine the correlation of performers (blind and independent) of angiography and echocardiography we will use the Kappa index.

The development of the risk model will be performed with logistic regression which dependent variable is the presence of MACE during hospitalization and 30 days (Wald method, backward). Variables for clinical and epidemiological history considered as relevant will be included, according also with the biological and epidemiological consistency and plausibility. The statistical criteria will be the inclusion of variables that in the bivariate analysis show p <0.20 and the exit criteria of the model will be p≥0.05.

The discriminative power of the model will be done with the area under the Receiver Operating Characteristic curve (ROC curve). The calibration will be done with the Hosmer-Lemeshow test. Relative risk with confidence intervals of 95 percent will be calculated. All hypothesis tests will be done under an alpha level of <0.05.

TIME OF DEVELOPMENT: Two years.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients of any gender between 18 and 90 years old
* Diagnosed with Acute Coronary Syndrome (STEMI/ NSTEMI/ Unstable angina - according to international diagnostic criteria - ACC / AHA / ESC)

Exclusion Criteria:

* Cardiomyopathies
* Congenital Disease
* Acute Pulmonary Embolism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of any gender between 18 and 90 years old, diagnosed with Acute Coronary Syndrome (STEMI/ NSTEMI/ Unstable angina - according to international diagnostic criteria - ACC / AHA / ESC), attended in representative hospitals of tertiary care in the IMSS will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 21827 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Major Cardiovascular Events (MACE) | up to 1 year
  Follow-up will be done during hospitalization and 30 days, time of most Major Cardiovascular Events presentation (MACE: Reinfarction, myocardial ischemia, heart failure, electrocardiographic complications and / or death ) derived from the timing of initial treatment or lack of it

SECONDARY OUTCOMES:
medical care cost in Instituto Mexicano del Seguro Social | 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Borrayo, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Gabriela Borrayo Sanchez, Mexico City, Mexico